CLINICAL TRIAL: NCT06452485
Title: Postoperative Re-irradiaTion With and Without HYPERthermia: Toxicity, Quality of Life and Survival in Patients With Locoregional Recurrent Breast Cancer
Acronym: RT-HYPE
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); Comprehensive Cancer Centre The Netherlands (Other); Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Desiree H.J.G.D. van den Bongard, MD Ph, Dr, Amsterdam UMC, location VUmc
Other Study IDs: 2012094
Record Dates: First submitted 2024-05-03; First posted 2024-06-11 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Locoregional Recurrence; Breast Cancer; Re-irradiation; Hyperthermia
MeSH Terms: conditions — Breast Neoplasms; Hyperthermia | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative re-irradiation with hyperthermia: Postoperative re-irradiation with hyperthermia in patients with locoregional recurrent breast cancer
  Interventions: Other: No interventions, patient-reported outcomes (PROMs) and toxicity will be collected in both groups.
- Postoperative re-irradiation without hyperthermia: Postoperative re-irradiation without hyperthermia in patients with locoregional recurrent breast cancer
  Interventions: Other: No interventions, patient-reported outcomes (PROMs) and toxicity will be collected in both groups.

INTERVENTIONS:
Other: No interventions, patient-reported outcomes (PROMs) and toxicity will be collected in both groups. — Patients will receive standard of care. Patients need to fill in questionnaires, these are additional interventions for the included subject. Questionnaires for patient-reported outcomes (PROMs) and toxicity will be filled in one week before treatment, one week before re-irradiation, one week and three months after re-irradiation, one, two and five years after surgery.

SUMMARY:
In the Netherlands, breast cancer patients with locoregional recurrence (LRR) and high-risk factors are treated with postoperative re-irradiation with or without hyperthermia. Retrospective studies showed that 3-year locoregional control after postoperative re-irradiation with hyperthermia was 68-83%, and severe toxicity in up to 40% of LRR patients. Unfortunately, no prospective (randomized) data are available on clinical outcomes. Consequently, variation exists in hyperthermia-treatment and re-irradiation schedules. Prospective real-world data on oncological outcomes, toxicity and quality of life is highly needed for shared decision-making between patients and professionals. These data will be used in the design of a future randomized trial comparing postoperative re-irradiation and hyperthermia-treatment in high-risk LRR patients.

DETAILED DESCRIPTION:
The optimal management of LRR breast cancer is multidisciplinary, and based on various prognostic risk factors and previous treatments. The surgical treatment of local recurrences is salvage mastectomy after previous breast-conserving therapy, or local excision after previous mastectomy. Regional treatment of tumor-positive lymph nodes consists of axillary radiotherapy and/or lymph node dissection. High-risk LRR patients have an indication for postoperative irradiation to improve locoregional control and disease-free survival. In previously irradiated high-risk LRR patients, postoperative re-irradiation is administered with or without hyperthermia in the Netherlands depending on the treating center and treating professional. Before the preoperative systemic treatment era, primary re-irradiation with hyperthermia was the evidence-based standard of care in high-risk unresectable LRR. Hyperthermia was used to increase the therapeutic efficacy of re-irradiation. The introduction of preoperative systemic therapy in 2010 resulted in more resectable high-risk LRRs. This resulted in postoperative re-irradiation instead of primary re-irradiation in LRR patients, including variation in the use of hyperthermia. There is no evidence-based standard of care regarding the combination of postoperative re-irradiation with or without hyperthermia in high-risk LRR patients. The major problem is that only retrospective data and no prospective (randomized) data is available on oncological outcomes (survival and recurrence) and toxicity following postoperative re-irradiation and hyperthermia. Consequently, there is a high need to assess oncological outcomes and toxicity of postoperative re-irradiation with or without hyperthermia in a randomized controlled trial (RCT). So far, an RCT has not been feasible due to the large variation in postoperative re-irradiation and hyperthermia, and preferences regarding hyperthermia-treatment by professionals. In the RT-HYPE study, the investigators evaluate oncological outcomes, toxicity and quality of life in high-risk LRR patients, including the harmonization of hyperthermia-treatment. The results of the RT-HYPE study are needed for the optimization of the shared decision making (SDM) process on post-operative re-irradiation with or without hyperthermia, between professionals and patients. In addition, these results allow to set-up a future RCT comparing postoperative re-irradiation with and without hyperthermia treatment.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance scale ≤2
* >=18 years
* Patients with a LRR breast cancer after postoperative irradiation of the primary breast cancer. LRR is defined as a local and/or regional recurrence, including patients with a second primary ipsilateral breast cancer.
* Patients treated with salvage mastectomy with high-risk* tumor characteristics or local excision with an indication for postoperative re-irradiation.
* Previously treated with whole or partial breast irradiation.
* (Neo)adjuvant systemic therapy (NST) is allowed.
* Use of (FES/FDG-)PET-CT in staging of nodal and disseminated disease.
* Oligometastases in lymph nodes in the mediastinum, neck, contralateral axillary/supraclavicular region (up to a maximal number of five) is allowed.
* Adequate communication and understanding skills of the Dutch language.

Exclusion Criteria:

* Diagnosed with primary breast sarcoma
* Have a low-risk LRR after previous breast-conserving surgery/therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older with an indication for postoperative re-irradiation with or without hyperthermia, eligible patients with a LRR with high-risk characteristics treated with mastectomy/local excision and postoperative re-irradiation, or mastectomy/local excision and postoperative re-irradiation with hyperthermia. Patients also treated with (neo-)adjuvant systemic treatment and/or with oligometastases (<=5 metastases), are allowed to be part of the study population.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Patient-reported toxicity according to PRO-CTCAE in LRR patients | Five years
  Patient-reported toxicity according to PRO-CTCAE after a median follow-up of five years after diagnosis of (subsequent) LRR disease.

SECONDARY OUTCOMES:
Quality of Life at 2 and 5 years after diagnosis of LRR disease | at 2 and 5 years after diagnosis of LRR disease
  EORTC-C30
Quality of Life at 2 and 5 years after diagnosis of LRR disease | at 2 and 5 years after diagnosis of LRR disease
  EORTC -BR45
LRR-free survival in LRR patients | at 2 and 5 years after diagnosis of LRR disease
distant metastasis-free survival in LRR patients | at 2 and 5 years after diagnosis of LRR disease
breast-cancer event-free survival in LRR patients | at 2 and 5 years after diagnosis of LRR disease
overall survival in LRR patients | at 2 and 5 years after diagnosis of LRR disease
Referral patterns in patients diagnosed with LRR | 5 year
  Referral patterns (per institute, professional, patient-related factors including performance status, and travel distance).

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Van Den Bongard, Dr, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided